CLINICAL TRIAL: NCT02855411
Title: A 12 Week, Phase 2, Randomized, Double-blind, Placebo Controlled, Parallel Group Study To Evaluate The Safety And Efficacy Of Pf-04958242 In Subjects With Cognitive Impairment Associated With Schizophrenia (CIAS)
Brief Title: A Study To Evaluate The Safety And Efficacy Of PF-04958242 In Subjects With Cognitive Impairment Associated With Schizophrenia (CIAS)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated prematurely Sept 22, 2016 following an internal portfolio prioritization. It is not due to any safety concern or change in benefit:risk assessment.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: B1701019; POC (Other: Alias Study Number)
Record Dates: First submitted 2016-07-27; First posted 2016-08-04 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Cognitive Impairment Associated With Schizophrenia (CIAS)
MeSH Terms: interventions — PF-04958242

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0.15 mg PF-04958242 (Experimental): Participants received 0.15 mg oral capsule, twice daily (BID) for 12 weeks
  Interventions: Drug: PF-04958242
- 0.5 mg PF-04958242 (Experimental): Participants received 0.5 mg oral capsule, twice daily (BID) for 12 weeks
  Interventions: Drug: PF-04958242
- Placebo (Placebo Comparator): Participants received matching placebo oral capsule, twice daily (BID) for 12 weeks
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: PF-04958242 — Administered as specified in the treatment arm
  Arms: 0.15 mg PF-04958242; 0.5 mg PF-04958242
Drug: placebo — placebo, twice daily (BID) for 12 weeks, capsule
  Other Names: Administered as specified in the treatment arm
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether PF-04958242 is safe and effective in the treatment of cognitive dysfunction in schizophrenia subjects

DETAILED DESCRIPTION:
This study was previously posted by Pfizer, Inc. Sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Otherwise healthy male and/or female subjects between the ages of 18 and 50 years, inclusive, with Diagnostic Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) diagnosis of schizophrenia of at least 2 years duration as confirmed by the M.I.N.I 7.0 for Psychotic Disorders
* Evidence of stable schizophrenia symptomatology >=3 months (ie, no hospitalizations for schizophrenia, no increase in level of psychiatric care due to worsening of symptoms of schizophrenia).
* Subjects must be in ongoing maintenance atypical antipsychotic therapy (except clozapine), on a stable treatment regimen for >=2 months prior to Baseline/Day 1, including concomitant psychotropic treatments. Subjects should be on no more than 2 background antipsychotics.
* Subject must have an identified informant
* Subject must reside in a stable living situation for at least 12 weeks prior to Screening.

Key Exclusion Criteria:

* Subjects with a current DSM-5 diagnosis of schizoaffective disorder in the judgment of the investigator.
* Subjects with a current DSM-5 diagnosis of major depressive episode, manic and hypomanic episode, panic disorder, agoraphobia, social anxiety disorder, obsessive-compulsive disorder, post-traumatic stress disorder, generalized anxiety disorder on the M.I.N.I 7.0 for Psychotic Disorders or in the judgment of the investigator.
* Subjects with a lifetime DSM-5 diagnosis of antisocial personality disorder, anorexia nervosa, bulimia nervosa, binge-eating disorder on the M.I.N.I 7.0 for Psychotic Disorders or in the judgment of the investigator.
* Subjects who meet the DSM-5 diagnosis of moderate or severe psychoactive substance use disorder (excluding nicotine dependence) within 12 months of screening on the M.I.N.I 7.0 for Psychotic Disorders interview and as determined by the investigator.
* Subjects with significant extrapyramidal symptoms which have not been stabilized with anticholinergics.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2016-09-26 (Actual); Study Completion 2016-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (16):
- United States (16):
  - Collaborative Neuroscience Network, LLC (Investigator Site File Location), Garden Grove, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Excell Research, Inc, Oceanside, California
  - NRC Research Institute, Orange, California
  - California Neuropsychopharmacology Clinical Research Institute, LLC (CNRI-San Diego, LLC), San Diego, California
  - Collaborative Neuroscience Network, LLC, Torrance, California
  - Atlanta Center For Medical Research, Atlanta, Georgia
  - Alexian Brothers Centers for Psychiatric Research, Hoffman Estates, Illinois
  - Chinmay K. Patel, D.O., Hoffman Estates, Illinois
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - CBH Health, LLC, Gaithersburg, Maryland
  - Hassman Research Institute, Berlin, New Jersey
  - CRI Worldwide, LLC, Marlton, New Jersey
  - Research Strategies of Memphis, LLC, Memphis, Tennessee
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Northwest Clinical Research Center, Bellevue, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 35 participants were screened before study termination.
Pre-assignment Details: No participants had been randomized to receive study drug or placebo before study termination.
Groups:
- Overall (PF-04958242/Placebo): Participants were to take PF-04958242 0.15 milligram (mg), or PF-04958242 0.5 mg, or the matched placebo twice daily (BID) for approximately 85 consecutive days, with the last dose taken in the morning on Day 85.
Period: Overall Study
Arm/Group | Overall (PF-04958242/Placebo)
Started | 35
Assigned to Study Treatment | 0
Completed | 0
Not Completed | 35
Not completed — Study terminated by sponsor | 21
Not completed — Does not meet entrance criteria | 14

BASELINE CHARACTERISTICS:
Population: A total of 35 participants were screened. Study was terminated before any participants were treated.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the MCCB (MATRICS Consensus Cognitive Battery) Working Memory Domain to Week 12
Description: The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (ie, working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). The MCCB yields scores for individual tests that assess specific cognitive domains as well as a composite score. Scores for the individual tests and the overall composite score for all tests are calculated according to the developers' recommended scoring algorithms.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

2. Primary Outcome: Change From Baseline in the UPSA-VIM (University of California, San Diego [UCSD] Performance Based Skills Assessment - Validation of Intermediate Measures) to Week 12
Description: The UPSA-VIM is a functional capacity measure of 5 general skills that were previously identified as essential to functioning in the community: general organization, finance, social/communications, transportation, and household chores. The UCSD Performance Based Skills Assessment involves role play tasks that are administered as simulations of events that the person might encounter in the community.
Time Frame: Baseline, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

3. Secondary Outcome: Scale for the Assessment and Rating of Ataxia (SARA)
Description: SARA is a clinical scale that is based on a semi--quantitative assessment of cerebellar ataxia on an impairment level and complements the brief neurological examination. The SARA has 8 items that are related to gait, stance, sitting, speech, finger-chase test, nose-finger test, fast alternating movements and heel-shin test.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Categorical Results on the Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS responses are mapped to the Columbia Classification Algorithm of Suicide Assessment (C-CASA). C-SSRS assesses whether participant experienced following: completed suicide (Category 1); suicide attempt (Category 2) (response of "Yes" on "actual attempt"); preparatory acts toward imminent suicidal behavior (Category 3) ("Yes" on "aborted attempt", or "interrupted attempt", or "preparatory acts or behavior"); suicidal ideation (Category 4) ("Yes" on "wish to be dead", or "non-specific active suicidal thoughts", or "active suicidal ideation with methods without intent to act or some intent to act, without specific plan or with specific plan and intent"); self-injurious behavior, no suicidal intent (Category 7) ("Yes" on "has participant engaged in non-suicidal self-injurious behavior"). Number of participants with "Yes" response for above mentioned categories was to be assessed.
Time Frame: Baseline, followed by weekly (Weeks 1 throughout 12), and 28 days after last dose
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline in the MCCB Neurocognitive Composite (Excluding Social Cognition Domain) to Week 12
Description: The MCCB is a cognitive battery to assess 7 domains recommended by the MATRICS initiative (ie, working memory, verbal learning, speed of processing, attention/vigilance, visual learning, social cognition, reasoning and problem solving). The MCCB yields scores for individual tests that assess specific cognitive domains as well as a composite score. Scores for the individual tests and the overall composite score for all tests are calculated according to the developers' recommended scoring algorithms. The MCCB neurocognitive score contains all of the tests and domains of the MCCB composite score with the exception of social cognition.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline in MCCB Overall Composite (Including All 7 Domains) to Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline in Each of the 6 Individual MCCB Domain Scores (Excluding MCCB Working Memory) to Week 12
Description: as for outcome 1
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline in the SCI-PANSS (Structured Clinical Interview Positive and Negative Symptoms Scale) Total to Week 12
Description: The SCI-PANSS includes 3 scales and 30 items: 7 items that make up the Positive Scale; 7 items that make up the Negative Scale; and 16 items that make up the General Psychopathology Scale. The sum of the 30 items is defined as the total score.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline in the SCI-PANSS Positive, Negative and General Psychopathology Subscales to Week 12
Description: The SCI--PANSS includes 3 scales and 30 items: 7 items that make up the Positive Scale; 7 items that make up the Negative Scale; and 16 items that make up the General Psychopathology Scale. The Subscale scores are the sum of corresponding individual items.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in the CGI-S (Clinical Global Impression-Severity) to Week 12
Description: The CGI--S consists of a single 7 point rating score of illness severity. Raters select 1 response based on the following question, "Considering your total clinical experience with this particular population, how mentally ill is your patient at this time?" Scores are: 1=Normal, not ill at all; 2=Borderline mentally ill; 3=Mildly ill; 4=Moderately ill; 5=Markedly ill; 6=Severely ill; or 7=Among the most severely ill participants.
Time Frame: Baseline, Week 2, Week 6, Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

11. Secondary Outcome: CGI-I (Clinical Global Impression-Improvement) at Week 12
Description: The CGI-I consists of a single 7 point rating score total improvement, regardless of whether or not the change is due entirely to drug treatment. Raters select 1 response based on the following question, "Compared to your patient's condition at the beginning of treatment, how much has your patient changed?" Scores are: 1=Very much improved; 2=Much improved; 3=Minimally improved; 4=No change; 5=Minimally worse; 6=Much worse; or 7=Very much worse. For the CGI-I, the participant's condition at the Day 1 (baseline) visit is the criterion for judging improvement at subsequent visits.
Time Frame: Week 12
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. AEs comprised both SAEs and non-SAEs. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. All AEs (serious and non-serious) occurring following start of treatment or increasing in severity in any period were to be considered as a treatment emergent AE.
Time Frame: For AEs, the time frame was from taking first dose through and including last visit (28 days after the last dose), up to 113 days. For SAEs, the time frame was from the time that the participant provided informed consent to last visit, up to 143 days.
Population: Study was terminated before participants were treated. No AE data was collected and there were no SAEs reported during the screening phase.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with laboratory test abnormalities without regard to baseline abnormality is assessed. Laboratory test parameters include hematology, clinical chemistry, urinalysis, follicle stimulating hormone, urine drug screen, and pregnancy test.
Time Frame: Screening up to Week 12 or early termination
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Electrocardiogram (ECG) Findings
Description: ECG criteria of potential clinical concern: 1) QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization): greater than or equal to (>=) 140 milliseconds (msec), >=50% increase from baseline; 2) PR interval (the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization): >=300 msec, >=25% increase when baseline is greater than (>) 200 msec or >=50% increase when baseline is less than or equal to (<=) 200 msec; 3) QTcF interval (time from ECG Q wave to the end of the T wave corresponding to electrical systole corrected using Fridericia's formula): absolute value of 450 to less than (<) 480 msec, 480 to <500 msec, >=500 msec; an increase from baseline of 30 to <60 msec or >=60 msec.
Time Frame: Screening up to Week 12 or early termination
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

15. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Findings
Description: Vital signs criteria of potential clinical concern: 1) systolic blood pressure <90 millimeters of mercury (mm Hg); 2) change from baseline of systolic blood pressure >=30 mm Hg; 3) diastolic blood pressure <50 mm Hg; 4) change from baseline of diastolic blood pressure >=20 mm Hg; 5) supine pulse rate <40 or >120 beats per minute (bpm); 6) standing pulse rate <40 or >140 bpm.
Time Frame: Screening up to Week 12 or early termination
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

16. Secondary Outcome: Number of Participants With Abnormalities in Neurological Examination
Description: The extended neurological examination includes observation for cerebellar (intention) tremor and for non-cerebellar tremors (eg, resting or positional), finger nose, heel shin, Romberg, tandem walking, positional and gaze-evoked nystagmus, reflexes, muscle strength, cranial nerves, sensory function of upper and lower extremities. The brief neurological examination includes an assessment of motor and sensory function, cranial nerves, reflexes, non-cerebellar tremor (eg, resting or positional) and cerebellar function. The assessment of cerebellar function is complemented by the Scale for the Assessment and Rating of Ataxia (SARA), a clinical scale based on a semi-quantitative assessment of cerebellar ataxia on an impairment level.
Time Frame: Screening up to Week 12 or early termination
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

17. Secondary Outcome: Number of Participants With Abnormalities in Physical Examination
Description: A full physical examination includes head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The brief physical examination is focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms.
Time Frame: Screening up to Week 12 or early termination
Population: Study was terminated before participants were treated and no data was collected for the endpoints.
Arm/Group | Overall (PF-04958242/Placebo)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: For SAEs, the time frame was from the time that the participant provided informed consent to last visit, up to 143 days. For AEs, the time frame was from taking first dose through and including last visit (28 days after the last dose), up to 113 days.
Description: Study was terminated before participants were treated. All the consented 35 participants were monitored/assessed for SAEs. No other (non-serious) AEs were collected/assessed because no participants were dosed.
Arm/Group | Overall (PF-04958242/Placebo)
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
This study was terminated due to Pfizer portfolio prioritization. No participants had been randomized to receive study drug or placebo. There is no safety or efficacy data to report for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.